CLINICAL TRIAL: NCT03430141
Title: Nutritarian Women's Health Study to Reduce Chronic Disease
Brief Title: A Nutritarian Study to Evaluate the Effectiveness of Lifestyle Changes in Chronic Disease Prevention, Especially Cancer
Acronym: NWHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Jay Sutliffe, Associate Professor, Northern Arizona University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nutritarian Women's Study
Record Dates: First submitted 2017-08-30; First posted 2018-02-12 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Chronic Disease; Cancer; Cardiovascular Diseases; Diabetes Mellitus; Lifestyle-related Condition; Mental Health Wellness 1; Sleep; Nutritional and Metabolic Disease; Nutrition Related Cancer; Nutritional Imbalance; Thyroid
MeSH Terms: conditions — Chronic Disease; Neoplasms; Cardiovascular Diseases; Diabetes Mellitus; Mental Disorders; Metabolic Diseases; Thyroid Diseases

STUDY DESIGN:
Intervention Model Description: Hybrid effectiveness-implementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention for all participants (Experimental): Nutritarian Diet-style: Intervention for all participants: All participants are exposed to the same nutrition treatment/intervention protocol.
  Interventions: Other: Nutritarian Diet-style

INTERVENTIONS:
Other: Nutritarian Diet-style — Nutritarian Diet-style: Daily consumption of greens, beans/legumes, a variety of other vegetables, fresh or frozen fruits, nuts, seeds and whole grains. Participants are encouraged to minimize consumption of refined grains, vegetable oils, processed foods, and to limit animal products.

SUMMARY:
The Nutritarian Women's Health Study (NWHS) is a long-term hybrid effectiveness-implementation study on the effect of the Nutritarian Diet on the occurrence, recurrence, and progression of chronic diseases (including all forms of cancer and cardiometabolic risk factors).

DETAILED DESCRIPTION:
The Nutritional Research Foundation, in conjunction with Northern Arizona University, is conducting a long-term health study for women ages 18 and older. This study will address the effects of a nutrient dense, plant-rich diet on the long-term risks of cancer and other chronic diseases.

Participants enroll in a 30-day training module which outlines the benefits of a nutrient-dense, plant-rich diet. At the conclusion of those videos and written modules, they take a short quiz to assess their knowledge and they can enroll in the full study.

All participation is online with ongoing modules on nutrition and lifestyle. There is a comprehensive health history and lifestyle index to be completed. Nutrition questionnaires will be administered an average of every 3-6 months; PHQ-9 (Patient Health Questionnaire) & PSQI (Pittsburgh Sleep Quality Index) questionnaires an average of every 12 months; serum cardiometabolic measures and liquid biopsies an average of every 18 months.

ELIGIBILITY:
Inclusion criteria:

* Women only
* Age 18 years and older.
* Must be willing to complete an online program
* Follow the dietary guidelines as outlined to the best of their ability.
* English-speaking
* US residents
* Have internet access
* Pregnant women are eligible

Exclusion criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 18 years and older
Enrollment: 2898 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Nutrition Intervention | Every 12 months, up to 10 years.
  Adherence to the recommended dietary protocol with the Nutritarian Health Indicator (©Joel Furhman MD). Scored by points (90-100 excellent, 80-89 good, 70-79 average, <69 poor).

SECONDARY OUTCOMES:
Weight Management | Every 12 months, up to 10 years.
  Height/weight/BMI of participants through self-reported measurements. Weight and height will be combined to report BMI in kg/m^2.
Waist Measurement | Every 12 months, up to 10 years.
  Self-measured and reported measurements in inches.
Hip Measurement | Every 12 months, up to 10 years.
  Self-measured and reported measurements in inches.
Mental Health | Every 12 months, up to 10 years.
  PHQ-9 (Patient Health Questionnaire-9). Tool designed for screening, diagnosing, monitoring and measuring the severity of depression. Scoring: 5-9 (minimal symptoms), 10-14 (minor depression, dysthymia, mild major depression), 15-19 (major depression, moderately severe), and >20 (major depression, severe).
Sleep quality assessment | Every 12 months, up to 10 years.
  PSQI (Pittsburgh Sleep Quality Index). Tool designed to evaluate sleep quality over a 1 month interval. Scoring 0-21 points. Any score >5 indicates sleep impairment, with higher scores designating poorer sleep and greater impact on daily life.
Cancer prevalence | Every 12 months, up to 10 years.
  Self-reported occurrence, recurrence, and progression of cancer at any site. Will be expressed as frequency distribution across the study population.
Chronic disease prevalence | Every 12 months, up to 10 years.
  Self-reported occurrence, recurrence, and progression of chronic disease (diabetes, cardiovascular disease, inflammatory disease). Will be expressed as frequency distribution across the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Sutliffe, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
We are considering making this data available to other researchers after we have a substantial number of participants enrolled.
Supporting Information: Study Protocol, CSR
Time Frame: Open October 31, 2016. Closed December 31. 2019.
Access Criteria: please contact study office at nwhs@nau.edu for information

REFERENCES:
- [Result] Sutliffe JT, Fuhrman JH, Carnot MJ, Beetham RM, Peddy MS. Nutrient-dense, Plant-rich Dietary Intervention Effective at Reducing Cardiovascular Disease Risk Factors for Worksites: A Pilot Study. Altern Ther Health Med. 2016 Sep;22(5):32-6. PMID 27622958
- [Result] Sarter B. Effect of a high nutrient density diet on long-term weight loss: a retrospective chart review. Altern Ther Health Med. 2011 Nov-Dec;17(6):10; author reply 10. No abstract available. PMID 22314713
- [Result] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Result] Yokoyama Y, Barnard ND, Levin SM, Watanabe M. Vegetarian diets and glycemic control in diabetes: a systematic review and meta-analysis. Cardiovasc Diagn Ther. 2014 Oct;4(5):373-82. doi: 10.3978/j.issn.2223-3652.2014.10.04. PMID 25414824
- [Result] Sutliffe JT, Wilson LD, de Heer HD, Foster RL, Carnot MJ. C-reactive protein response to a vegan lifestyle intervention. Complement Ther Med. 2015 Feb;23(1):32-7. doi: 10.1016/j.ctim.2014.11.001. Epub 2014 Dec 3. PMID 25637150
- [Result] Fuhrman J, Sarter B, Glaser D, Acocella S. Changing perceptions of hunger on a high nutrient density diet. Nutr J. 2010 Nov 7;9:51. doi: 10.1186/1475-2891-9-51. PMID 21054899
- [Result] Gonzales JF, Barnard ND, Jenkins DJ, Lanou AJ, Davis B, Saxe G, Levin S. Applying the precautionary principle to nutrition and cancer. J Am Coll Nutr. 2014;33(3):239-46. doi: 10.1080/07315724.2013.866527. Epub 2014 May 28. PMID 24870117
- [Result] Tucker KL, Hallfrisch J, Qiao N, Muller D, Andres R, Fleg JL; Baltimore Longitudinal Study of Aging. The combination of high fruit and vegetable and low saturated fat intakes is more protective against mortality in aging men than is either alone: the Baltimore Longitudinal Study of Aging. J Nutr. 2005 Mar;135(3):556-61. doi: 10.1093/jn/135.3.556. PMID 15735093